CLINICAL TRIAL: NCT01897233
Title: A Phase 3, Open-label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Lumacaftor in Combination With Ivacaftor in Subjects 6 Through 11 Years of Age With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Brief Title: Study of Lumacaftor in Combination With Ivacaftor in Subjects 6 Through 11 Years of Age With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX13-809-011
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lumacaftor/Ivacaftor (LUM/IVA) (Experimental): Part A Cohort 1: Participants aged 6 through 8 years will receive LUM 200 milligram (mg) in fixed-dose combination with IVA 250 mg orally every 12 hours (q12h) for 14 days.
  Part A Cohort 2: Participants aged 9 through 11 years will receive LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 14 days.
  Part B: Participants aged 6 through 11 years will receive LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 24 weeks.
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor

INTERVENTIONS:
Drug: Lumacaftor
  Other Names: VX-809
Drug: Ivacaftor
  Other Names: VX-770

SUMMARY:
This is a Phase 3, 2-part (Part A and Part B), open-label, multicenter study to evaluate the pharmacokinetics, safety, and tolerability of lumacaftor in combination with ivacaftor in subjects with cystic fibrosis aged 6 to 11 years who have the F508del-mutation in the cystic fibrosis transmembrane conductance regulator (CFTR) gene.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF defined as: with 2 CF-causing mutations, chronic sinopulmonary disease or gastrointestinal/nutritional abnormalities
* Subjects who weigh ≥15 kg without shoes at Screening Visit
* Subjects who are homozygous for the F508del-CFTR mutation
* Subjects with percent predicted forced expiratory volume in 1 second (FEV1) of 70% to 105% (inclusive) (Part A) or ≥40% (Part B) at Screening Visit where the predicted values are adjusted for age, sex, and height using the Wang equation
* Subjects with stable CF disease and who are willing to remain on stable CF medication regimen
* Able to swallow tablets

Exclusion Criteria:

* History of any illness or condition that might confound the results of the study or pose an additional risk in administering study drug to the subject
* Acute respiratory infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 28 days before Day 1 of the study
* Abnormal liver function as defined in the protocol at Screening Visit
* Abnormal renal function as defined in the protocol at Screening Visit
* History of solid organ or hematological transplantation
* Ongoing participation in an investigational drug study or prior participation in an investigational drug study within 30 days prior of Screening Visit
* History or evidence of lens opacity or cataract at Screening Visit
* Colonization with organisms associated with a more rapid decline in pulmonary status at Screening Visit (Part A only)
* A standard 12-lead ECG demonstrating QTcF >450 msec at Screening Visit

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (19):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Long Beach, California
  - Palo Alto, California
  - Aurora, Colorado
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Kansas City, Missouri
  - St Louis, Missouri
  - Buffalo, New York
  - Rochester, New York
  - Syracuse, New York
  - Charleston, South Carolina
  - Austin, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Toronto, Ontario, Canada

REFERENCES:
- [Background] Wang X, Dockery DW, Wypij D, Fay ME, Ferris BG Jr. Pulmonary function between 6 and 18 years of age. Pediatr Pulmonol. 1993 Feb;15(2):75-88. doi: 10.1002/ppul.1950150204. PMID 8474788
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Milla CE, Ratjen F, Marigowda G, Liu F, Waltz D, Rosenfeld M; VX13-809-011 Part B Investigator Group *. Lumacaftor/Ivacaftor in Patients Aged 6-11 Years with Cystic Fibrosis and Homozygous for F508del-CFTR. Am J Respir Crit Care Med. 2017 Apr 1;195(7):912-920. doi: 10.1164/rccm.201608-1754OC. PMID 27805836

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 2 parts - Part A and Part B. Part A consisted of 2 cohorts, in which participants aged 6 to 8 years were enrolled in Cohort 1 and participants aged 9 to 11 years were enrolled in Cohort 2. Part B consisted of a single cohort. Participants from Part A may have also participated in Part B of the study.
Groups:
- Lumacaftor/Ivacaftor (LUM/IVA): Part A Cohort 1: Participants aged 6 through 8 years received LUM 200 milligram (mg) in fixed-dose combination with IVA 250 mg orally every 12 hours (q12h) for 14 days.
  Part A Cohort 2: Participants aged 9 through 11 years received LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 14 days.
  Part B: Participants aged 6 through 11 years received LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 24 weeks.
Period: Part A (14 Days)
Arm/Group | Lumacaftor/Ivacaftor (LUM/IVA)
Started | 10
Part A Cohort 1 (6 to 8 Years) | 5
Part A Cohort 2 (9 to 11 Years) | 5
Completed | 10
Not Completed | 0
Period: Part B (24 Weeks)
Arm/Group | Lumacaftor/Ivacaftor (LUM/IVA)
Started | 58 (6 participants from Part A also participated in Part B of the study.)
Completed | 54
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who received at least 1 dose of study drug.
Groups:
- Lumacaftor/Ivacaftor (LUM/IVA): Part A Cohort 1: Participants aged 6 through 8 years received LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 14 days.
  Part A Cohort 2: Participants aged 9 through 11 years received LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 14 days.
  Part B: Participants aged 6 through 11 years received LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 24 weeks.
Arm/Group | Lumacaftor/Ivacaftor (LUM/IVA)
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] — Data were planned to be reported separately for Part A and Part B of the study. Here "n" signifies participants who were evaluable for specified part of the study.
  years
    Part A Cohort 1 (n=5) | 6.6 (0.89)
    Part A Cohort 2 (n=5) | 9.6 (0.89)
    Part B (n=58) | 9.1 (1.53)
Sex/Gender, Customized [Number; unit: participants] — Data were planned to be reported separately for Part A and Part B of the study. Here "n" signifies participants who were evaluable for specified part of the study.
  participants
    Part A Cohort 1 (n=5): Female | 1
    Part A Cohort 1 (n=5): Male | 4
    Part A Cohort 2 (n=5): Female | 1
    Part A Cohort 2 (n=5): Male | 4
    Part B (n=58): Female | 31
    Part B (n=58): Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Part A: Observed Plasma Concentration of Lumacaftor (LUM) and Ivacaftor (IVA) at Hour 4 Post-dose (C4h) on Day 1
Time Frame: 4 hours post-morning dose on Day 1
Population: The Pharmacokinetic (PK) Set included all enrolled participants who received the study drug and for whom the primary PK data were considered to be sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part A Overall Arm: LUM/IVA: All participants aged 6 through 11 years who received LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 14 days.
Arm/Group | Part A Overall Arm: LUM/IVA
Number analyzed (Participants) | 10
nanogram per milliliter (ng/mL)
  LUM | 15200 (6740)
  IVA | 1920 (727)

2. Primary Outcome: Part A: Observed Plasma Concentration of Lumacaftor (LUM) and Ivacaftor (IVA) at Hour 4 Post-dose (C4h) on Day 14
Time Frame: 4 hours post-morning dose on Day 14
Population: The PK Set included all enrolled participants who received the study drug and for whom the primary PK data were considered to be sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A Overall Arm: LUM/IVA
Number analyzed (Participants) | 10
ng/mL
  LUM | 24500 (10400)
  IVA | 622 (322)

3. Primary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time 0 to End of Dosing Interval (AUCtau) of Lumacaftor (LUM) and Ivacaftor (IVA)
Description: The AUCtau is the area under the concentration versus time curve from time 0 to time tau, where tau is the time at the end of dosing interval.
Time Frame: Day 14 (pre-morning dose, 4, 6, 12, and 24 hours post-morning dose for LUM; pre-morning dose, 2, 4, 6, 12 hours post-morning dose for IVA)
Population: as for outcome 2
Measure: Median (Full Range); unit: ng*hr/mL
Arm/Group | Part A Overall Arm: LUM/IVA
Number analyzed (Participants) | 10
ng*hr/mL
  LUM | 387600 [280700 to 640800]
  IVA | 6838 [2689 to 12100]

4. Primary Outcome: Part B: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, inpatient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. AEs with start date or increased severity on or after the first study drug dose to Week 26 were considered treatment-emergent.
Time Frame: Day 1 up to Week 26
Population: The Safety Set included all participants who received any amount of Part B study drug
Measure: Number; unit: participants
Groups:
- Part B: LUM/IVA: Participants aged 6 through 11 years received LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 24 weeks.
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 58
participants
  AEs | 55
  SAEs | 4

5. Secondary Outcome: Part A: Observed Plasma Concentration of Lumacaftor Metabolite (M28-LUM) and Ivacaftor Metabolites (M1-IVA and M6-IVA) at Hour 4 Post-dose (C4h) on Day 1 and 14
Time Frame: Day 1, Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A Overall Arm: LUM/IVA
Number analyzed (Participants) | 10
ng/mL
  M28-LUM (Day 1) | 176 (79.0)
  M1-IVA (Day 1) | 3940 (1380)
  M6-IVA (Day 1) | 1810 (981)
  M28-LUM (Day 14) | 2040 (1230)
  M1-IVA (Day 14) | 2380 (1360)
  M6-IVA (Day 14) | 4240 (1990)

6. Secondary Outcome: Part A: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, inpatient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. AEs with start date or increased severity on or after the first study drug dose through the end of Part A were considered treatment-emergent.
Time Frame: Day 1 up to Day 28
Population: The Safety Set included all participants who received at least 1 dose of study drug. Here "n" signifies those subjects who were evaluable for the specified cohort.
Measure: Number; unit: participants
Arm/Group | Part A Overall Arm: LUM/IVA
Number analyzed (Participants) | 10
participants
  Part A Cohort 1: AEs (n=5) | 4
  Part A Cohort 1: SAEs (n=5) | 0
  Part A Cohort 2: AEs (n=5) | 3
  Part A Cohort 2: SAEs (n=5) | 0

7. Secondary Outcome: Part B: Average Absolute Change From Baseline in Sweat Chloride at Day 15 and at Week 4
Description: Sweat samples were collected using an approved collection device. Baseline was defined as the average of the measurements at screening and on Day 1 pre-dose. Average of Day 15 and Week 4 measurements was taken and change was calculated as: Average (Day 15 and Week 4 measurement) minus Baseline measurement.
Time Frame: Baseline, Day 15 and Week 4
Population: The Full Analysis Set (FAS) included all Part B enrolled participants who were exposed to any amount of Part B study drug. Here "Number of Participants" analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 57
millimole per liter (mmol/L) | -19.7 [-23.2 to -16.3]

8. Secondary Outcome: Part B: Absolute Change in Sweat Chloride From Week 24 at Week 26
Description: Sweat samples were collected using an approved collection device. Change = Week 26 minus Week 24.
Time Frame: Week 24, Week 26
Population: The FAS included all Part B enrolled participants who were exposed to any amount of Part B study drug. Here "Number of Participants" analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 47
mmol/L | 21.3 [18.6 to 24.0]

9. Secondary Outcome: Part B: Absolute Change From Baseline in Body Mass Index (BMI) at Week 24
Description: BMI was defined as weight in kilogram (kg) divided by height*height in square meter (m^2).
Time Frame: Baseline, Week 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram per square meter (kg/m^2)
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 56
kilogram per square meter (kg/m^2) | 0.64 [0.46 to 0.83]

10. Secondary Outcome: Part B: Absolute Change From Baseline in BMI-for-age Z-score at Week 24
Description: BMI was defined as weight in kg divided by height*height in m^2. z-score is a statistical measure to evaluate how a single data point compares to a standard. It describes whether a mean was above or below the standard and how unusual the measurement is, with range from -infinity to +infinity; where 0: same mean, >0: a greater mean, and <0: a lesser mean than the standard. BMI, adjusted for age and sex, was analyzed as BMI-for-age z-score (BMI z-score). The BMI-for-age z-scores were calculated using National Center for Health Statistics growth charts.
Time Frame: Baseline, Week 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 56
z-score | 0.15 [0.08 to 0.22]

11. Secondary Outcome: Part B: Absolute Change From Baseline in Weight at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms (kg)
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 56
kilograms (kg) | 2.6 [2.2 to 3.0]

12. Secondary Outcome: Part B: Absolute Change From Baseline in Weight-for-age Z-score at Week 24
Description: Z-score is a statistical measure to evaluate how a single data point compares to a standard. It describes whether a mean was above or below the standard and how unusual the measurement is, with range from -infinity to +infinity; where 0: same mean, >0: a greater mean, and <0: a lesser mean than the standard. Weight, adjusted for age and sex, was analyzed as weight-for-age z-score (weight z-score). The weight-for-age z-scores were calculated using National Center for Health Statistics growth charts.
Time Frame: Baseline, Week 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 56
z-score | 0.13 [0.07 to 0.19]

13. Secondary Outcome: Part B: Absolute Change From Baseline in Height at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeter (cm)
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 56
centimeter (cm) | 2.9 [2.6 to 3.2]

14. Secondary Outcome: Part B: Absolute Change From Baseline in Height-for-age Z-score at Week 24
Description: Z-score is a statistical measure to evaluate how a single data point compares to a standard. It describes whether a mean was above or below the standard and how unusual the measurement is, with range from -infinity to +infinity; where 0: same mean, >0: a greater mean, and <0: a lesser mean than the standard. Height, adjusted for age and sex, was analyzed as height-for-age z-score (height z-score). The height-for-age z-scores were calculated using National Center for Health Statistics growth charts.
Time Frame: Baseline, Week 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 56
z-score | 0.03 [-0.02 to 0.09]

15. Secondary Outcome: Part B: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score at Week 24
Description: The CFQ-R is a validated patient-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Baseline, Week 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 56
Units on a scale | 5.4 [1.4 to 9.4]

16. Secondary Outcome: Part B: Absolute Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) Domains at Week 24
Description: The TSQM is a 14-item self-administered questionnaire which measures participants' experiences with their medication on four dimensions: effectiveness, side effects, convenience and global satisfaction. For each dimension, responses are added and transformed to a scale from 0 to 100, where higher scores indicate greater satisfaction.
Time Frame: Baseline, Week 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 50
units on a scale
  Change at Week 24: Effectiveness | 9.2 [4.3 to 14.1]
  Change at Week 24: Side Effects | -0.3 [-1.4 to 0.8]
  Change at Week 24: Convenience | 11.1 [7.1 to 15.1]
  Change at Week 24: Global Score | 3.6 [-2.0 to 9.1]

17. Secondary Outcome: Part B: Pre-dose Concentration (Ctrough) and 3 to 6 Hours Post-dose Concentration (C3-6hr) of Lumacaftor, Lumacaftor Metabolite (M28-LUM), Ivacaftor and Ivacaftor Metabolites (M1-IVA and M6-IVA)
Description: Ctrough and C3-6hr for lumacaftor, M28 lumacaftor (lumacaftor metabolite), ivacaftor, M1 ivacaftor (ivacaftor metabolite), and M6 ivacaftor (ivacaftor metabolite) were calculated. Ctrough was observed pre-dose concentration. C3-6hr was observed concentration at 3 to 6 hours post- dose.
Time Frame: For Ctrough: pre-morning dose on Week 4, Week 6 and Week 24; For C3-6hr: 3 to 6 hours post-morning dose on Day 1, 15 and Week 4
Population: The PK Set included all enrolled participants who received the study drug and for whom the primary PK data were considered to be sufficient and interpretable. Here "n" signifies those participants who were evaluable at the specified time point for the given category.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B: LUM/IVA
Number analyzed (Participants) | 58
ng/mL
  C3-6h LUM (Day 1) (n=57) | 17100 (6260)
  C3-6h IVA (Day 1) (n=57) | 1980 (850)
  C3-6h M28-LUM (Day 1) (n=57) | 186 (96.3)
  C3-6h M1-IVA (Day 1) (n=57) | 4170 (1940)
  C3-6h M6-IVA (Day 1) (n=57) | 2040 (1650)
  C3-6h LUM (Day 15) (n=55) | 21400 (6850)
  C3-6h IVA (Day 15) (n=55) | 751 (433)
  C3-6h M28-LUM (Day 15) (n=55) | 1660 (843)
  C3-6h M1-IVA (Day 15) (n=55) | 2670 (1330)
  C3-6h M6-IVA (Day 15) (n=55) | 4360 (2340)
  C3-6h LUM (Week 4) (n=54) | 22000 (8470)
  C3-6h IVA (Week 4) (n=54) | 779 (389)
  C3-6h M28-LUM (Week 4) (n=54) | 1730 (884)
  C3-6h M1-IVA (Week 4) (n=54) | 2800 (1410)
  C3-6h M6-IVA (Week 4) (n=54) | 4690 (3360)
  Ctrough LUM (Week 4) (n=53) | 12300 (6780)
  Ctrough IVA (Week 4) (n=53) | 171 (228)
  Ctrough M28-LUM (Week 4) (n=53) | 1780 (903)
  Ctrough M1-IVA (Week 4) (n=53) | 684 (816)
  Ctrough M6-IVA (Week 4) (n=53) | 2490 (2150)
  Ctrough LUM (Week 16) (n=53) | 11500 (6020)
  Ctrough IVA (Week 16) (n=52) | 153 (150)
  Ctrough M28-LUM (Week 16) (n=53) | 1610 (859)
  Ctrough M1-IVA (Week 16) (n=53) | 690 (627)
  Ctrough M6-IVA (Week 16) (n=53) | 2360 (1570)
  Ctrough LUM (Week 24) (n=51) | 11400 (5300)
  Ctrough IVA (Week 24) (n=51) | 118 (87.2)
  Ctrough M28-LUM (Week 24) (n=51) | 1710 (947)
  Ctrough M1-IVA (Week 24) (n=51) | 493 (409)
  Ctrough M6-IVA (Week 24) (n=51) | 1790 (1180)

ADVERSE EVENTS:
Time Frame: Part A: Day 1 up to Day 28; Part B: Day 1 up to Week 26
Description: For Part A: MedDRA 16.0 and For Part B: MedDRA 18.1 was used.
Groups:
- Part A Cohort 1: LUM/IVA: Participants aged 6 through 8 years received LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 14 days.
- Part A Cohort 2: LUM/IVA: Participants aged 9 through 11 years received LUM 200 mg in fixed-dose combination with IVA 250 mg orally q12h for 14 days.
Arm/Group | Part A Cohort 1: LUM/IVA | Part A Cohort 2: LUM/IVA | Part B: LUM/IVA
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 4/58
Other Adverse Events (participants affected / at risk) | 4/5 | 3/5 | 55/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Cohort 1: LUM/IVA (N=5) | Part A Cohort 2: LUM/IVA (N=5) | Part B: LUM/IVA (N=58)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Cohort 1: LUM/IVA (N=5) | Part A Cohort 2: LUM/IVA (N=5) | Part B: LUM/IVA (N=58)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 29
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 12
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 12
Dizziness (Nervous system disorders) | 0 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 8
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 6
Nausea (Gastrointestinal disorders) | 0 | 0 | 6
Vomiting (Gastrointestinal disorders) | 0 | 0 | 6
Constipation (Gastrointestinal disorders) | 1 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2
Faecal volume increased (Gastrointestinal disorders) | 0 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3
Pulmonary function test decreased (Investigations) | 0 | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1
Blood creatinine decreased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1
Crystal urine present (Investigations) | 0 | 0 | 1
Eosinophil count decreased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1
Pseudomonas test positive (Investigations) | 0 | 0 | 1
Streptococcus test positive (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Forced Expiratory Volume Decreased (Investigations) | 0 | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 6
Pyrexia (General disorders) | 1 | 0 | 6
Application site erythema (General disorders) | 0 | 0 | 2
Application site urticaria (General disorders) | 0 | 0 | 2
Application site vesicles (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Vessel puncture site reaction (General disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 11
Otitis media (Infections and infestations) | 0 | 0 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2
Otitis externa (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Abscess limb (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3
Seasonal allergy (Immune system disorders) | 0 | 0 | 3
House dust allergy (Immune system disorders) | 0 | 0 | 1
Mycotic allergy (Immune system disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 2
Cataract (Eye disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Enuresis (Renal and urinary disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to limited sampling and instances of missing data, C4h was reported instead of Cmax as an approximation of maximum concentration. Sparse PK sampling scheme was optimized around parent compounds which limited the estimation of AUC for metabolites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.